CLINICAL TRIAL: NCT02958995
Title: Epidemiologic Study Of Diabetes And Cancer Risk
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: AD-4833_403B; EUPAS10335 (Registry Identifier: EU PAS)
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2, Cancer
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full KPNC Cohort: Participants who were members of the KPNC registry (with or without diabetes) were followed up to 15 years (1997-2011) in this epidemiological study.
  Interventions: Other: No Intervention
- Survey Responders: A subset of KPNC members who completed the Kaiser Diabetes Registry Survey in 1994-1996 and among a random sample of KPNC members who completed the Member Health Survey (MHS), in 1996, 1999, 2002, or 2005 were followed up to 15 years (1997-2011) in this epidemiological study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study was to evaluate whether treatment with pioglitazone is associated with risk of incident cancer at the 10 most common sites in a cohort of participants with recognized diabetes along with the assessment of association between diabetes severity and cancer risk.

DETAILED DESCRIPTION:
The study enroll a large population of approximately 252467 participants. This epidemiology study of diabetes and cancer risk is an expansion study which would include estimation of cancer rate among KPNC members with or without diabetes and the relative risks of cancers associated with a diagnosis of diabetes. The study included diabetes participants who were KPNC members between 1997 and 2011. It also included a subset of participants who took the 1996/7 diabetes survey and Member Health Survey (MHS) in 1993, 1999, 2001 or 2003.

This multi-center trial was conducted in the United States of America. The overall time to participate in this study was approximately 15.5 years. The participants were followed-up from January 1, 1997 up to December 31, 2011.

ELIGIBILITY:
Inclusion Criteria: 1. has been in the KPNC diabetes registry Diabetes Mellitus (DM) registry, aged 40 years or older and are members of KPNC as of January 1, 1997 and had no prior diagnosis of the cancer of interest.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a historical diagnosis of Type 2 diabetes mellitus (T2DM) with pioglitazone exposure identified from the Kaiser Permanente of Northern California(KPNC) Diabetes Registry (with or without diabetes) and had completed Member Health Survey (MHS) were enrolled in the epidemiology study.
Sampling Method: Probability Sample
Enrollment: 2738161 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- See also: Interim Results Report — https://www.takeda.com/siteassets/en-us/home/external-reference/clinicaltrials.gov/ad-4833-403-fum_35.4_kpnc_interim_results_report-2011-12-07.pdf
- See also: 10 Yr Study Report — https://www.takeda.com/siteassets/en-us/home/external-reference/clinicaltrials.gov/ad4833-403_kpnc_10_common_cancers_10-yr_study_report.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 01 July 1997 to 30 June 2011.
Pre-assignment Details: Participants with a historical diagnosis of Type 2 diabetes mellitus (T2DM) with pioglitazone exposure identified from the Kaiser Permanente of Northern California(KPNC) Diabetes Registry (with or without diabetes) and had completed Member Health Survey (MHS) were enrolled in the epidemiology study.
Groups:
- Survey Responders Cohort: A subset of KPNC members who completed the Kaiser Diabetes Registry Survey in 1994-1996 and among a random sample of KPNC members who completed the Member Health Survey (MHS), in 1996, 1999, 2002, or 2005 were followed up to 15 years (1997-2011) in this epidemiological study.
Period: Overall Study
Arm/Group | Full KPNC Cohort | Survey Responders Cohort
Started | 2630666 | 107495
Completed | 2630666 | 107495
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The observational study population consisted of T2DM participants who were identified from KPNC registry (with or without diabetes) and had completed the KPNC survey and MHS in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full KPNC Cohort | Survey Responders Cohort | Total
Number analyzed (Participants) | 2630666 | 107495 | 2738161
Age, Customized [Number; unit: participants]
  40 - 49 years | 1501084 (11.6) | 30256 (12.9) | 1531340
  50 - 59 years | 570636 | 24585 | 595221
  60 - 69 years | 322517 | 25582 | 348099
  70 - 79 years | 170136 | 22028 | 192164
  greater than or equal to (>=) 80 years | 66293 | 5044 | 71337
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1353782 | 54418 | 1408200
  Male | 1276884 | 53077 | 1329961
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1339805 | 67837 | 1407642
  Black | 171604 | 10167 | 181771
  Hispanic | 322046 | 11871 | 333917
  Asian or Pacific Islander | 312730 | 13508 | 326238
  Other | 87901 | 2728 | 90629
  Unknown | 396580 | 1384 | 397964

OUTCOME MEASURES:

1. Primary Outcome: Age and Sex-Standardized Incidence Rates for the 10 Most Common Cancers Stratified by Diabetes Status
Description: Age and gender adjusted incidence rates, stratified by diabetes status, was calculated using the direct method (2000 US Census as standard), with further stratification on calendar year. Cancer incidence rates were calculated with attention to the proper allocation of at-risk person-time. The association between diabetes and risk of each of the 10 most common cancers was assessed using Cox proportional hazards regression models with control for available potential confounders: age, gender. Similarly, Cox regression technique was used to examine the association between diabetes status and cancer risk among survey responders with adjustment for additional potential confounding variable.
Time Frame: 15 years
Population: Analysis population included participants from KPNC registry (with or without diabetes) and had completed the MHS in the epidemiology study.
Measure: Number (95% Confidence Interval); unit: Incidence per 100,000 person-years
Arm/Group | Full KPNC Cohort | Survey Responders Cohort
Number analyzed (Participants) | 2630666 | 107495
Incidence per 100,000 person-years
  Prostate, Diabetes Status: No | 380.2 [375.6 to 384.9] | 421.9 [393.6 to 450.2]
  Prostate, Diabetes Status: Yes | 308.0 [299 to 316.9] | 281.9 [265.7 to 298.2]
  Female Breast, Diabetes Status: No | 291.8 [288.2 to 295.5] | 310.7 [287.6 to 333.8]
  Female Breast, Diabetes Status: Yes | 286.9 [276.3 to 297.5] | 287.9 [266.1 to 309.6]
  Lung/Bronchus, Diabetes Status: No | 111.3 [109.7 to 113.0] | 116.1 [107.0 to 125.3]
  Lung/Bronchus, Diabetes Status: Yes | 108.8 [104.9 to 112.6] | 105.9 [98.5 to 113.2]
  Colon, Diabetes Status: No | 69.1 [67.8 to 70.5] | 75.5 [67.9 to 83.1]
  Colon, Diabetes Status: Yes | 93.5 [89.7 to 97.3] | 97.3 [90.1 to 104.5]
  Non-Hodgkin lymphoma, Diabetes: No | 39.5 [38.5 to 40.5] | 40.6 [34.6 to 46.6]
  Non-Hodgkin lymphoma, Diabetes: Yes | 45.6 [42.8 to 48.4] | 43.2 [37.7 to 48.6]
  Corpus uteri, Diabetes Status: No | 55.9 [54.3 to 57.5] | 59.7 [49.6 to 69.8]
  Corpus uteri, Diabetes Status: Yes | 112.1 [104.9 to 119.2] | 106.2 [92.7 to 119.6]
  Pancreas, Diabetes Status: No | 18.8 [18.1 to 19.5] | 18.5 [14.9 to 22.1]
  Pancreas, Diabetes Status: Yes | 47.3 [44.6 to 49.9] | 37.1 [32.3 to 41.9]
  Kidney/Renal Pelvis, Diabetes Status: No | 23.5 [22.7 to 24.2] | 21.5 [17.2 to 25.7]
  Kidney/Renal Pelvis, Diabetes Status: Yes | 39.5 [36.8 to 42.2] | 34.5 [29.0 to 40.0]
  Rectal, Diabetes Status: No | 24.6 [23.8 to 25.4] | 26.7 [21.7 to 31.7]
  Rectal, Diabetes Status: Yes | 31.1 [28.7 to 33.4] | 31.9 [26.6 to 37.2]
  Melanoma, Diabetes Status: No | 42.5 [41.5 to 43.5] | 55.8 [48.5 to 63.0]
  Melanoma, Diabetes Status: Yes | 30.6 [28.2 to 32.9] | 31.7 [26.8 to 36.7]

2. Primary Outcome: Hazard Ratio for Risk of 10 Common Cancers Associated With Diabetes
Description: The association between diabetes and risk of each of the 10 most common cancers was assessed by calculating hazard ratio using Cox proportional hazards regression models with control for available potential confounders: age, gender and calendar years. Cox regression techniques was used to examine the association between DM status and cancer risk with adjustment for potential confounding variables in the survey respondent cohort.
Time Frame: 15 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Full KPNC Cohort | Survey Responders Cohort
Number analyzed (Participants) | 2630666 | 107495
Ratio
  Prostate, Diabetes Status | 0.81 [0.78 to 0.83] | 0.77 [0.68 to 0.86]
  Female Breast, Diabetes Status | 1.01 [0.98 to 1.05] | 0.98 [0.86 to 1.12]
  Lung/Bronchus, Diabetes Status | 0.99 [0.96 to 1.03] | 0.84 [0.74 to 0.96]
  Colon, Diabetes Status | 1.36 [1.31 to 1.42] | 1.18 [1.01 to 1.38]
  Non-Hodgkin lymphoma, Diabetes | 1.14 [1.07 to 1.21] | 1.06 [0.85 to 1.33]
  Corpus uteri, Diabetes Status | 1.82 [1.71 to 1.95] | 1.67 [1.28 to 2.18]
  Pancreas, Diabetes Status | 2.50 [2.35 to 2.67] | 2.38 [1.78 to 3.18]
  Kidney/Renal Pelvis, Diabetes Status | 1.56 [1.46 to 1.67] | 1.37 [1.04 to 1.82]
  Rectal, Diabetes Status | 1.25 [1.16 to 1.35] | 1.41 [1.05 to 1.89]
  Melanoma, Diabetes Status | 0.73 [0.68 to 0.79] | 0.69 [0.55 to 0.86]

ADVERSE EVENTS:
Description: Due to the observational nature of study individual adverse events (AEs) were not planned to be collected and reported.
Arm/Group | Full KPNC Cohort | Survey Responders Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.